CLINICAL TRIAL: NCT05788419
Title: A Sonographic Study of the Hip Joints in Ice Hockey League Players
Brief Title: Sonographic Study of Hip Joint in Hockey Players
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Malá Jitka, Clinical Professor, Charles University, Czech Republic
Other Study IDs: Hybner, sonography
Record Dates: First submitted 2023-03-01; First posted 2023-03-28 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Hip Joint Contracture
Keywords: hockey; hip joint; sonography
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- examination group: Group of active hockey players
  Interventions: Diagnostic Test: sonography
- control group: Group of athletes, non hockey players
  Interventions: Diagnostic Test: sonography

INTERVENTIONS:
Diagnostic Test: sonography — imaging method, functional test of hip joint
  Other Names: FADIR test

SUMMARY:
The aim is to determine whether the game of ice hockey has an effect on structural changes in the hip joint. The parameter to be investigated will be the increased frequency of structural changes of the hip joint in ice hockey players compared to a control group. Participants in the study will undergo MSK sonographic examination of both hip joints followed by functional hip mobility testing. The functional testing consists of three tests. Data will be processed in MS Office in MS Word, and the resulting data will be subject to statistical evaluation.

DETAILED DESCRIPTION:
The examined hip joint structure will be examined monographically and simultaneously using functional tests, the Patrick test, a passive test of the range of motion in the hip joint to external and internal rotation in the joint, FADDIR test. Approximately 20 probands will be enrolled in the study based on voluntary participation from a group of players of the Charles University hockey team Prague, who have a valid medical examination with no restrictions on eligibility for selected sporting activities. The second group will consist of approximately 20 additional probands from the U20 age group of ice hockey players enrolled voluntarily with a valid medical examination with no restrictions on eligibility for the selected sporting activities. In addition, approximately 20 volunteers of the same age range will be included in the study and form the control group. In total, there will be approximately 60 participants in the study.

The conditions for inclusion in the first and second test groups will be an age range of 19-28 years, playing ice hockey for 6 years at least three times a week in the standard training regime of Czech ice hockey clubs. The player must be a registered player, i.e. his/her health condition must be suitable for ice hockey. The exclusion criteria for the test group will be persons outside the defined age limit with acute or chronic illnesses for any reason and persons with post-traumatic hip and pelvic conditions.

The inclusion criteria for the third control group will be the same age range of 19-28 years and no acute, especially infectious, diseases and persons with post-traumatic hip and pelvic conditions. This will be a normal recreational sporting population with no registration affiliation in any sport.

ELIGIBILITY:
Inclusion Criteria:

* a valid medical examination with no restrictions on eligibility for selected sports activities
* playing ice hockey from the age of 6 at least three times a week in the standard training regime of Czech ice hockey clubs
* registered player, i.e. his/her health must be fit to play ice hockey.

Exclusion Criteria:

* persons outside the defined age limit
* with acute or chronic illnesses for any reason
* persons with post-traumatic hip and pelvic conditions

Ages: 19 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Twenty probands will be included in the study based on voluntary participation from the group of players of the university hockey team UK hockey Prague; the second group will consist of another 20 probands from the age group U20 ice hockey players included in the basis of voluntary participation, who have a valid medical examination without restrictions on eligibility for selected sports activities. In addition, approximately 20 volunteers of the same age range will be included in the study and form the control group. In total, there will be approximately 60 participants in the study.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
sonography picture identification | 20 min
  identification of a higher prevalence of structural changes of the hip joint in hockey players

SECONDARY OUTCOMES:
comparison of the functional tests | 20 min
  Determining whether functional tests correlate with sonographic findings

CONTACTS AND LOCATIONS:
Overall Officials: Jitka Malá, Dr, Principal Investigator — Charles University Prague, Czech Republic
Locations (1):
- Charles University, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Undecided